CLINICAL TRIAL: NCT00416195
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Explore the Safety And Tolerability of Doses of E2007 up to a Maximum of 12 mg In Patients With Refractory Partial Seizures
Brief Title: Exploring the Safety And Tolerability of Doses of E2007 up to a Maximum of 12 mg In Patients With Refractory Partial Seizures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Collaborators: Eisai Limited (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-G000-208; 2006-003702-26 (EudraCT Number)
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Results first posted 2012-11-22 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2013-08

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- E2007 (Experimental): 2 mg E2007 once daily for 2 weeks (Days 1 to 14), then 4 mg E2007 once daily for 2 weeks (Days 15 to 28), then 6 mg E2007 once daily for 2 weeks (Days 29 to 42), then 8 mg E2007 once daily for 2 weeks (Days 43 to 56), then 10 mg E2007 once daily for 2 weeks (Days 57 to 70), then 12 mg E2007 once daily for 6 weeks (Days 71 to 112).
  Interventions: Drug: E2007
- Placebo (Placebo Comparator): Matching placebo once daily for 16 weeks (Days 1 to 112)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2007
  Arms: E2007
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel group study to determine the maximum tolerated dose of E2007. Epilepsy patients with refractory partial seizures will be divided into two groups of 24 patients each. One group will be patients who take concomitant inducing AEDs (anti-epileptic drugs) and the second group will be patients who do not take concomitant inducing AEDs. In each group, 18 patients will receive E2007 (dose escalating to a maximum of 12 mg per day) and six will receive placebo.

ELIGIBILITY:
INCLUSION CRITERIA

1. Provide written informed consent signed by patient or legal guardian prior to entering the study or undergoing any study procedures.
2. Are reliable and willing to make themselves available for the study period and are able to record seizures and report AEs themselves or have a caregiver who can record and report the events.
3. Male and female patients will be eligible for enrollment. Females should be either of nonchildbearing potential as a result of surgery or menopause (1 year after onset), or of childbearing potential and practicing a medically acceptable method of contraception (e.g., abstinence, a barrier method plus spermicide, or intrauterine device [IUD]) for at least 1 month before Visit 1 (Screening) and for 1 month after the end of the study. They must also have a negative serum beta-human chorionic gonadotropin (B-hCG) at Screening. Those females using hormonal contraceptives must also be using an additional approved method of contraception (e.g., a barrier method plus spermicide or IUD) starting with the Baseline Phase and continuing throughout the entire study period.
4. Are between the ages of 18 and 70 years of age, inclusive.
5. Are of 40 kg (88 pounds) of weight or more.
6. Have the diagnosis of epilepsy with partial seizures with or without secondarily generalized seizures according with the International League Against Epilepsy's Classification of Epileptic Seizures (1981). Diagnosis should have been established by clinical history, electroencephalogram and computed tomography/magnetic resonance imaging of the brain performed within the last 10 years and consistent with localization-related epilepsy.
7. Have uncontrolled partial seizures despite having been treated with at least three different AEDs (given concurrently or sequentially) for at least 2 years.
8. Have averaged at least three partial seizures per month, with no 21-day seizure-free period during the 2 months preceding randomization. This should be documented in the form of medical history, medical records, or photocopied records of the patient diary/patient chart. Simple partial seizures without motor signs will not be counted towards this inclusion criterion.
9. Are currently being treated with one to three (maximum) marketed and approved AEDs and are known to take their medications as directed. Use of a vagal nerve stimulator is not considered an AED by this criterion.
10. Are on a stable dose of the same AEDs for the 1 month prior to Visit 1.
11. If using a vagal nerve stimulator, it must have been implanted at least 5 months prior to Visit 1. Stimulator parameters may not be changed for at least 1 month prior to Visit 1 or during the study. Magnet use will be allowed and documented throughout the study.

EXCLUSION CRITERIA

1. Have participated in a study involving administration of an investigational compound within 3 months of Visit 1 (Screening), or within 5 half-lives of the previous investigational compound, whichever is longer, or who have been previously treated with E2007.
2. Presence of nonmotor simple partial seizures only.
3. Presence of primary generalized epilepsies or seizures, such as absences, myoclonic epilepsies, Lennox-Gastaut syndrome.
4. History of status epilepticus in the past year or seizure clusters where individual seizures cannot be counted.
5. Show evidence of clinically significant disease (cardiac, respiratory, gastrointestinal, renal disease, etc) that, in the opinion of the investigator, could affect either the patient's safety or the conduct of the study.
6. Show evidence of significant, active, hepatic disease. Stable elevations of liver enzymes, alanine aminotransferase (ALT), and aspartate aminotransferase (AST) due to concomitant medications will be allowed if they are less than 2 times the ULN.
7. Show evidence of significant active hematological disease such as a white blood cell (WBC) count <= 2500/µL (2.50 1E+09/L), an absolute neutrophil count <= 1000/µL (1.00 1E+09/L), or a platelet count <100,000/mm^3.
8. Patients with clinically significant ECG abnormality, including prolonged QTc (defined as QTc >=450 msec using Fridericia's correction).
9. Presence of major active psychiatric disease. Patients taking a stable dose of selective serotonin reuptake inhibitor antidepressant (except fluvoxamine) will be allowed.
10. Presence of a progressive central nervous system (CNS) disease, including degenerative CNS diseases and progressive tumors.
11. Have a history of psychogenic seizures in the past 2 years.
12. Pregnant or lactating females.
13. Have a history of drug abuse in the past 2 years and/or positive finding on urinary drug screening, other than prescribed medication.
14. Have a history of alcohol abuse in the past 2 years, and/or positive finding on urinary drug screen.
15. Have had multiple drug allergies (dermatological, hematological, or organ toxicity) or one or more severe drug reactions.
16. Allergy to lactose.
17. Concomitant use of felbamate or use of felbamate within 2 months prior to Visit 1.
18. Concomitant use or use within the 4 weeks prior to Visit 1 of neuroleptics, monoamine oxidase (MAO) inhibitors, barbiturates (except for seizure control indication), benzodiazepines (other than occasional intermittent use), and narcotic analgesics.
19. Frequent need of rescue benzodiazepines (two or more times a month).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Yang, MD, MBA, Study Director — Eisai Inc.
Locations (2):
- Latvia (2):
  - P. Stradina Clinical University Hospital, Riga
  - Hospital Gailezers, Riga

REFERENCES:
- [Derived] Bresnahan R, Hill RA, Wang J. Perampanel add-on for drug-resistant focal epilepsy. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD010961. doi: 10.1002/14651858.CD010961.pub2. PMID 37059702
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920

RESULTS

PARTICIPANT FLOW:
Groups:
- Perampanel: 2 mg perampanel once daily for 2 weeks (Days 1 to 14), then 4 mg perampanel once daily for 2 weeks (Days 15 to 28), then 6 mg perampanel once daily for 2 weeks (Days 29 to 42), then 8 mg perampanel once daily for 2 weeks (Days 43 to 56), then 10 mg perampanel once daily for 2 weeks (Days 57 to 70), then 12 mg perampanel once daily for 6 weeks (the last 2 weeks of the Titration Phase [Days 71 to 84] and a 4-week Maintenance Phase [Days 85 to 112])
Period: Overall Study
Arm/Group | Placebo | Perampanel
Started | 10 | 38
Completed | 8 | 34
Not Completed | 2 | 4
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 1
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Perampanel | Total
Number analyzed (Participants) | 10 | 38 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.5 (12.05) | 40.7 (11.99) | 43.1 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 20 | 25
  Male | 5 | 18 | 23
Race/Ethnicity, Customized [Number; unit: participants] — Race
  participants
    Caucasian | 10 | 38 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders During the Maintenance Phase
Description: A patient is a responder if she/he experiences a 50% or greater reduction in seizure frequency from the baseline phase.
Time Frame: Day 85 through Day 112
Population: ITT population- all subjects in the Safety Population (all randomized subjects who took at least 1 dose of study drug) who had at least 2 weeks of baseline seizure frequency data and at least 1 week of seizure frequency data after baseline (LOCF - last observation carried forward)
Measure: Number; unit: Percentage of Participants
Arm/Group | Placebo | Perampanel
Number analyzed (Participants) | 9 | 38
Percentage of Participants
  Responders (Yes) | 44.4 | 34.2
  Non-Responders (No) | 55.6 | 65.8

2. Secondary Outcome: Percentage Change in the 28-day Seizure Frequency From Baseline in the Maintenance LOCF
Time Frame: Baseline, Day 85 through Day 112
Population: ITT population (LOCF)
Measure: Median (Full Range); unit: Percent change
Arm/Group | Placebo | Perampanel
Number analyzed (Participants) | 9 | 38
Percent change | -46.4 [-81.5 to 221.0] | -35.4 [-100.0 to 93.3]

ADVERSE EVENTS:
Arm/Group | Placebo | Perampanel
Serious Adverse Events (participants affected / at risk) | 1/10 | 1/38
Other Adverse Events (participants affected / at risk) | 7/10 | 15/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Perampanel (N=38)
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Convulsions (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=10) | Perampanel (N=38)
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Rhinitis (Infections and infestations) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 6
Headache (Nervous system disorders) | 1 | 1
Muscle contractions involuntary (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No